CLINICAL TRIAL: NCT07096778
Title: A Phase II, Open-Label, Multicenter Study of Inobrodib in Combination With Pomalidomide and Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Inobrodib, Pomalidomide and Dexamethasone in Relapsed or Refractory Multiple Myeloma
Acronym: DoMMino-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CellCentric Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCS1477-04; 1012518 (Other: IRAS)
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma Refractory; Multiple Myeloma in Relapse
Keywords: Inobrodib; Pomalidomide; Pomalyst; Imnovid; Dexamethasone; p300-CBP Transcription Factors
MeSH Terms: interventions — pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Inobrodib in combination with pomalidomide and dexamethasone (Experimental)
  Interventions: Drug: Inobrodib; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Inobrodib — 20 mg orally twice daily (b.i.d.) 4 days on / 3 days off for each 28-day cycle.
  Other Names: CS1477
Drug: Pomalidomide — 4 mg orally once daily on Day 1 to 21 of each 28-day cycle
  Other Names: Pomalyst; Imnovid
Drug: Dexamethasone — 40 mg orally once daily on Days 1, 8, 15 and 22 for each 28-day cycle

SUMMARY:
The purpose of this study is to learn more about the anti-cancer activity of inobrodib, when given in combination with pomalidomide and dexamethasone, in patients with multiple myeloma that has come back following treatment and which no longer responds to available therapies. The study treatment will not be compared to any other treatment and patients will know what treatment they are receiving. This study will also further explore the side effects of inobrodib in combination with these other medicines.

DETAILED DESCRIPTION:
This is a Phase II, open-label, multicenter study to evaluate the efficacy and safety of inobrodib in combination with pomalidomide and dexamethasone (InoPd) in patients with relapsed and refractory multiple myeloma (RRMM).

Patients must be 18 years or older and be refractory to least one proteosome inhibitor (PI), one anti-CD38 monoclonal antibody (mAb) and pomalidomide. Patients must also be previously treated with an approved bispecific T-cell engager [TCE].

Approximately 100 patients will be treated with 20 mg of inobrodib administered orally twice daily (b.i.d.) 4 days on / 3 days off for each 28-day cycle. Pomalidomide and dexamethasone will be administered as per standard of care (SoC), i.e., with a starting dose of 4 mg orally once daily on Day 1 to 21 of each 28-day cycle for pomalidomide, and 40 mg orally once daily on Days 1, 8, 15 and 22 for each 28-day cycle for dexamethasone. Study treatment should be continued until disease progression, initiation of new anticancer therapy, unacceptable toxicity or the patient meets any criteria for withdrawal from the study.

The primary objective is to assess the efficacy of InoPd in terms of objective response rate (ORR) based on International Myeloma Working Group (IMWG) criteria and assessed by Independent Review Committee (IRC).

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age
* Prior diagnosis of MM as defined according to IMWG criteria and relapsed or refractory to the last line of therapy
* Eastern Co-operative Oncology Group (ECOG) performance status of 0 to 2
* Adequate hematological, renal and hepatic function
* Willingness to use highly effective contraceptive measures (if sexually active) with all sexual partners

Exclusion Criteria:

* Use of any investigational agent, chemotherapy, immunotherapy or anticancer agent from a previous clinical study within 14 days or 5 half-lives of first dose of study treatment, whichever is shortest; any antibody based therapy within 30 days
* Prior treatment with p300/CBP bromodomain inhibitors
* Known or suspected severe allergies to any active or inactive ingredients in the study medications (inobrodib, pomalidomide, dexamethasone) or any prior immunomodulatory drug (lenalidomide, thalidomide)
* Treatment with medicines or herbal supplements or foods (e.g. strong CYP3A4 inducers or inhibitors) that would interfere with treatment
* Major surgery within 4 weeks of the first dose of study treatment
* Live vaccine within 4 weeks of study treatment
* Active or unresolved adverse events
* Active malignancies (progressing or requiring change in treatment) in the last 24 months other than multiple myeloma
* Female patients who are pregnant or breast-feeding at any time during the study
* Any illness or medical history that would impact safety or compliance with study requirements or impact ability to interpret study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-22 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate, defined as the percentage of patients with a confirmed partial response (PR) or better, based on IMWG criteria and assessed by Independent Review Committee (IRC) | Assessed from enrollment to date of progressive disease or death from any cause, until the end of study (up to 48 months)

SECONDARY OUTCOMES:
ORR, defined as the percentage of patients with a confirmed PR or better, based on IMWG criteria assessed by Investigator | Assessed from enrollment to date of progressive disease or death from any cause, until the end of study (up to 48 months)
Duration of Response (DoR), defined as the duration of overall response by investigator and ICR | Assessed from enrollment to date of progressive disease or death from any cause, until the end of study (up to 48 months)
Time to Response (TTR), defined as time to confirmed PR or better, by investigator and ICR | Assessed from enrollment to date of progressive disease or death from any cause, until the end of study (up to 48 months)
Very Good Partial Response (VGPR) or better rate, defined as the percentage of patients with a confirmed VGPR or better, based on IMWG criteria and assessed by investigator and ICR | Assessed from enrollment to date of progressive disease or death from any cause, until the end of study (up to 48 months)
Complete Response (CR) or better rate, defined as the percentage of patients with a confirmed CR or better, based on IMWG criteria and assessed by investigator and ICR | Assessed from enrollment to date of progressive disease or death from any cause, until the end of study (up to 48 months)
Progression Free Survival (PFS), defined as the time from enrolment until the earliest date of Progressive Disease (PD), or death due to any cause, and assessed by investigator and ICR | Assessed from enrollment to date of progressive disease or death from any cause, until the end of study (up to 48 months)
Overall Survival (OS), defined as the time from enrolment to the date of death due to any cause | Assessed from enrollment to date of death from any cause, until the end of study (up to 48 months)
Incidence of treatment-emergent adverse events (TEAEs), vital signs and laboratory abnormalities | Assessed from start of treatment until 28 days after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Naseer Qayum, Study Director — CellCentric Ltd.
Locations (2):
- United Kingdom (2):
  - Royal Marsden NHS Foundation Trust, Sutton, London
  - Imperial College Healthcare NHS Trust, Hammersmith Hospital, London

IPD SHARING:
Plan to Share IPD: No
The final clinical study report will be provided to the Investigators. The Sponsor will publicly disclose study results through posting on ClinicalTrials.gov and any other applicable public registries in accordance with local regulations.